CLINICAL TRIAL: NCT01677728
Title: A Randomized, Controlled Trial of Target Therapy Plus Chemotherapy in Patients Undergoing Liver Resection for Colorectal Liver Metastases
Brief Title: Effect of Target Therapy on Patients Undergoing Synchronic Hepatectomy for Colorectal Liver Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Zhongshan hospital, Fudan University
Organization: Fudan University (Other)
Other Study IDs: ZSTCC; Xjianmin (Registry Identifier: Xjianmin)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer; Liver Tumor
Keywords: colorectal liver metastases; chemotherapy; cetuximab; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- arm A: patients received chemotherapy alone
- arm B: patients received target therapy combined with chemotherapy

SUMMARY:
The aim of this study is to explore whether target therapy in combination with chemotherapy as treatment could improve survival or tumor response in patients undergoing Synchronic Hepatectomy for Colorectal Liver Metastases.

DETAILED DESCRIPTION:
In patients with colorectal cancer (CRC), the liver is the most common site of hematogenous metastases. Approximately half of patients develop hepatic metastases during the course of the disease, and hepatic metastases are responsible for death in at least two thirds of CRC patients.

Over the past decade, due to the introduction of irinotecan-based or oxaliplatin-based combination chemotherapy, the median survival among patients with colorectal liver metastases (CLM) has increased from 6 ~8 months to more than 20 months5.In recent years, target therapy has rapidly gained attention for the treatment of CLM and is under active investigation.

Although numerous publications have reported the efficacy of target therapy in combination treatment for CLM patients, most of these studies focused solely on those patients without undergoing resection of liver metastases. In contrast, little work has concentrated on exploring the effection of target therapy for CLM patients undergoing Synchronic Hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 75 years old
* Performance status (ECOG) 0~1
* colorectal adenocarcinoma pathologically
* without any chemotherapy or radiotherapy
* liver metastases undergoing radical resection
* colorectal cancer undergoing radical resection
* no other metastases
* suitable for chemotherapy
* agreed by patients

Exclusion Criteria:

* age below 18 years old or greater than 75 years old
* haven't pathological diagnosis of colorectal adenocarcinoma with liver metastase
* with any chemotherapy or radiotherapy
* with other metastasis
* unresectable colorectal cancer or liver metastases
* unsuitable for chemotherapy or target therapy
* not agreed by patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From Zhongshan hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianmin, MD, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China